CLINICAL TRIAL: NCT06773338
Title: Does Playing Tetris Prevent the Development of Post-Traumatic Stress Disorder or Related Anxiety and Depressive Symptoms During and After Migration?
Brief Title: The Impact of Playing Tetris on Migrants' Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Collaborators: Stichting tot steun VCVGZ (Other)
Responsible Party: Principal Investigator, Mario Braakman, Professor, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLS_RP1253; IC2024-1 (Other Grant/Funding Number: Tilburg University Fund); 300.6700 3613 (Other Grant/Funding Number: Stichting tot Steun VCVGZ); 305.6700 3614 (Other Grant/Funding Number: Stichting tot Steun VCVGZ)
Record Dates: First submitted 2024-12-19; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Post-traumatic Stress Disorder (PTSD); Anxiety Symptoms; Depression Symptoms
Keywords: Post-traumatic stress disorder; PTSD; Anxiety; Depression; Refugees; Asylum seekers; Migrants; Tetris; Longitudinal
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment tetris group (Other): Randomly selected participants who reply to mental health and migration-related difficulties questionnaires are asked to play Tetris during the research.
  Interventions: Behavioral: Tetris
- Control group (Other): Randomly selected participants who reply to mental health and migration-related difficulties questionnaires, but do not play Tetris during the research.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Tetris — Randomly selected participants (migrants) are asked to play Tetris for at least 15 minutes on several occasions. These participants are asked while playing Tetris to try and remember bad events that recently happened to them. The participants play the classic version of the Tetris game directly on their mobile phone.
  Arms: Treatment tetris group
Other: No intervention — Participants do not receive any intervention.
  Arms: Control group

SUMMARY:
This study examines if playing Tetris prevents the development of Post-traumatic stress disorder or related anxiety and depressive symptoms. The investigators recruit 300 participants in total in Greece and in the Netherlands. The participants are immigrants who have applied for asylum at any point in the past. The participants are asked to answer three questionnaires (on Post-traumatic stress disorder, related anxiety and depressive symptoms, and post-migration living difficulties) on a recurring basis - once every 4 weeks, 12 times in total. Half of the participants (treatment group) are randomly selected to play Tetris after completing the questionnaires. Participants in the treatment group are instructed to play Tetris for at least 15 minutes while trying to remember bad things that recently happened to them. Tetris is administered at three instances and participants in the treatment group are encouraged to play Tetris in case of experiencing any traumatic events or having any intrusive memories during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Arabic-speaking immigrants of any gender who have applied for asylum in Greece or in the Netherlands, regardless of the outcome of their asylum application and their current residency status (rejected asylum seekers, recognized refugees, undocumented migrants).

Exclusion Criteria:

* Minors (under the age of 18).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic stress disorder | From enrolment to the end of the study (40 weeks)
  The investigators use the Primary Care Post-Traumatic Stress Disorder Screen for Diagnostic and Statistical Manual of Mental Disorders fifth edition (PC-PTSD-5)
Anxiety and depression symptoms | From enrolment to the end of the study (40 weeks)
  The investigators use the Kessler Psychological Distress Scale

SECONDARY OUTCOMES:
Post-migration living difficulties | From enrolment to the end of the study (40 weeks)
  In the course of the study, the investigators measure variation in post-migration living difficulties such as separation from family, social isolation, language barriers, etc. Participants are presented a checklist of items and asked to identify for each item if it has been a problem for them over the last month, with 4 possible answers for each item: 1) not a problem; 2) minor problem; 3) serious problem; 4) very serious problem.
  In addition, participants are asked if over the last month they have 1) been victimised in any way ; 2) had any negative experiences involving bureaucratic personnel or state officials; 3) had experiences that made them feel happy and gave them hope for the future (open questions).

CONTACTS AND LOCATIONS:
Locations (2):
- Upinion (online), The Hague, NL, Greece
- Upinion/the humanity Hub, The Hague, NL, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Tilburg University's standards and considering the sensitivity of the data collected from asylum seekers, the availability for reuse of the data will be subject to careful consideration and protection of privacy. The availability of the data for reuse will be determined on a case-by-case basis, taking into consideration the consent obtained from participants, any legal or ethical restrictions, and the level of identifiability of the data. To protect the privacy and confidentiality of the asylum seekers, data sharing will be done in a controlled manner.The availability of the data for reuse will be determined on a case-by-case basis, taking into consideration the consent obtained from participants, any legal or ethical restrictions, and the level of identifiability of the data.